CLINICAL TRIAL: NCT05082701
Title: Sentinel™ Trial: A Prospective Study Evaluating the Performance and Clinical Benefit of Personalized ctDNA-based MRD Testing to Detect Recurrence and Monitor Treatment Response in Patients With Solid Tumors
Acronym: Sentinel
Status: Terminated | Type: Observational
Why Stopped: Sentinel MRD test offers no additional or increased benefits to patients compared to current marketed alternatives
Sponsor: Strata Oncology (Industry)
Responsible Party: Sponsor
Other Study IDs: STR-005-001
Record Dates: First submitted 2021-09-09; First posted 2021-10-19 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples With DNA — 1. FFPE tumor tissue sample (study initiation collection)
  2. 20mL blood sample (collection every 3 months)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Sentinel™ Trial is a non-randomized, large-scale observational trial designed to: 1) evaluate the ability of circulating tumor DNA (ctDNA)-based minimal residual disease (MRD) testing to detect recurrence in advance of standard-of-care techniques across solid tumors, and 2) determine the clinical benefit of therapy in ctDNA-positive participants.

The study offers the opportunity to 1) serially monitor participants for ctDNA changes, 2) define ctDNA kinetics across tumor and therapy types, 3) identify participants with ctDNA evidence of MRD, and 4) understand the clinical benefit of ctDNA status on treatment outcomes.

DETAILED DESCRIPTION:
Patients with a confirmed diagnosis of a stage I through III solid tumor who have had definitive therapy or curative surgery within the last 5 years or are planning curative surgery may be eligible for the Sentinel Trial. Patients must have a surplus formalin-fixed paraffin-embedded tumor specimen available at screening, or a planned resection within 28 days of screening. To support ctDNA assessment, study procedures will be limited to serial blood draws repeated every 12 weeks until investigator determined recurrence. Upon recurrence, participants will remain on study for 3 years in survival follow-up.

ELIGIBILITY:
Study participants must meet all the inclusion criteria below to enroll:

1. Male or female participants ≥ 18 years of age;
2. Confirmed diagnosis of a stage 1-3 solid tumor;
3. Curative surgery or definitive therapy (e.g., chemoradiation, stereotactic body radiation therapy [SBRT]) completed <5 years ago without any current evidence of radiographical or biochemical recurrence, or planned within 28 days of consent;
4. Surplus formalin fixed paraffin embedded tumor specimen available;
5. Able to tolerate venipuncture for blood draws;
6. Primary diagnosis is not glioma or CNS disease;
7. Both the tumor tissue sample and blood sample pass the quantity and quality parameters to allow for a successful MRD test result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants must meet all the inclusion criteria listed to enroll; 1. Male or female participants ≥ 18 years of age; 2. Confirmed diagnosis of a stage 1-3 solid tumor; 3. Curative surgery or definitive therapy (e.g., chemoradiation, stereotactic body radiation therapy [SBRT]) completed <5 years ago without any current evidence of radiographical or biochemical recurrence, or planned within 28 days of consent; 4. Surplus formalin fixed paraffin embedded tumor specimen available; 5. Able to tolerate venipuncture for blood draws; 6. Primary diagnosis is not glioma or CNS disease; 7. Both the tumor tissue sample and blood sample pass the quantity and quality parameters to allow for a successful MRD test result.
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 8 years
  Evaluate ability of ctDNA-based MRD monitoring to detect disease recurrence in advance of SOC recurrence monitoring across solid tumors, as stratified by tumor type and adjuvant therapy status. With sensitivity being the proportion of participants with radiographic recurrence who first had a ctDNA recurrence and specificity being the proportion of participants without radiographic recurrence who did not first have a ctDNA recurrence.
ctDNA Response Rate | 8 years
  Determine the clinical benefit of treatment in ctDNA-positive participants, as stratified by therapy class (targeted, immuno-, chemo-, etc.), individual therapy, tumor type, stage, and biomarker status. With ctDNA response rate being the proportion of participants with >50% reduction in mean variant allele frequency (VAF) on-treatment at 3 months compared to baseline VAF.

SECONDARY OUTCOMES:
Disease Free Survival (DFS): Duration of time between initiation of treatment and radiographic recurrence (investigator assessment) or death | 8 years
  Determine the relationship between ctDNA response, clearance, and kinetics and radiographically determined disease-free survival and overall survival overall and as stratified by therapy class (targeted, immuno-, chemo-, etc.), individual therapy, tumor type, stage, and biomarker status.
Disease Free Survival (DFS): Duration of time between initiation of treatment and radiographic recurrence (investigator assessment) or death | 8 years
  Determine the clinical benefit of therapy versus surveillance in ctDNA-positive participants as stratified by therapy class (targeted, immuno-, chemo-, etc.), individual therapy, tumor type, and biomarker status (DFS, OS). With Disease Free Survival (DFS) being the duration of time between initiation of treatment and radiographic recurrence (investigator assessment) or death and Overall survival (OS) being the duration of time between initiation of treatment and death.
Disease Free Survival (DFS): Duration of time between initiation of treatment and radiographic recurrence (investigator assessment) or death | 8 years
  Determine the adjuvant therapy utilization rate stratified by ctDNA status, tumor type and tumor stage.

OTHER OUTCOMES:
Examine the interaction of baseline tissue derived biomarkers identified by StrataMRD testing with ctDNA status and kinetics | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Kat Kwiatkowski, PhD, Study Director — Strata Oncology
Locations (4):
- United States (4):
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Miller KD, Nogueira L, Mariotto AB, Rowland JH, Yabroff KR, Alfano CM, Jemal A, Kramer JL, Siegel RL. Cancer treatment and survivorship statistics, 2019. CA Cancer J Clin. 2019 Sep;69(5):363-385. doi: 10.3322/caac.21565. Epub 2019 Jun 11. PMID 31184787
- [Background] Bockelman C, Engelmann BE, Kaprio T, Hansen TF, Glimelius B. Risk of recurrence in patients with colon cancer stage II and III: a systematic review and meta-analysis of recent literature. Acta Oncol. 2015 Jan;54(1):5-16. doi: 10.3109/0284186X.2014.975839. Epub 2014 Nov 28. PMID 25430983
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Background] Coombes RC, Page K, Salari R, Hastings RK, Armstrong A, Ahmed S, Ali S, Cleator S, Kenny L, Stebbing J, Rutherford M, Sethi H, Boydell A, Swenerton R, Fernandez-Garcia D, Gleason KLT, Goddard K, Guttery DS, Assaf ZJ, Wu HT, Natarajan P, Moore DA, Primrose L, Dashner S, Tin AS, Balcioglu M, Srinivasan R, Shchegrova SV, Olson A, Hafez D, Billings P, Aleshin A, Rehman F, Toghill BJ, Hills A, Louie MC, Lin CJ, Zimmermann BG, Shaw JA. Personalized Detection of Circulating Tumor DNA Antedates Breast Cancer Metastatic Recurrence. Clin Cancer Res. 2019 Jul 15;25(14):4255-4263. doi: 10.1158/1078-0432.CCR-18-3663. Epub 2019 Apr 16. PMID 30992300
- [Background] Wu YL, Tsuboi M, He J, John T, Grohe C, Majem M, Goldman JW, Laktionov K, Kim SW, Kato T, Vu HV, Lu S, Lee KY, Akewanlop C, Yu CJ, de Marinis F, Bonanno L, Domine M, Shepherd FA, Zeng L, Hodge R, Atasoy A, Rukazenkov Y, Herbst RS; ADAURA Investigators. Osimertinib in Resected EGFR-Mutated Non-Small-Cell Lung Cancer. N Engl J Med. 2020 Oct 29;383(18):1711-1723. doi: 10.1056/NEJMoa2027071. Epub 2020 Sep 19. PMID 32955177
- [Background] Vidal J, Casadevall D, Bellosillo B, Pericay C, Garcia-Carbonero R, Losa F, Layos L, Alonso V, Capdevila J, Gallego J, Vera R, Salud A, Martin-Richard M, Nogue M, Cillan E, Maurel J, Faull I, Raymond V, Fernandez-Martos C, Montagut C. Clinical Impact of Presurgery Circulating Tumor DNA after Total Neoadjuvant Treatment in Locally Advanced Rectal Cancer: A Biomarker Study from the GEMCAD 1402 Trial. Clin Cancer Res. 2021 May 15;27(10):2890-2898. doi: 10.1158/1078-0432.CCR-20-4769. Epub 2021 Mar 16. PMID 33727257
- [Background] Powels, T.B. et al., Clinical outcomes in post-operative ctDNA-positive muscle-invasive urothelial carcinoma (MIUC) patients after atezolizumab adjuvant therapy. Annals of Oncology, 2020. 31(suppl_7): S1417-S1424.